CLINICAL TRIAL: NCT06286891
Title: Evaluation of Frailty, Physical Capacity and Lung Function in Postoperative Pulmonary Endarterectomy Patients: an Observational and Prospective Clinical Study
Brief Title: Frailty, Physical Capacity and Lung Function in Postoperative Pulmonary Endarterectomy Patients
Status: Recruiting | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Rafael M. Ianotti, PT, Clinical Research Coordinator - Physiotherapy Division - Heart Institute (InCor), University of Sao Paulo General Hospital
Other Study IDs: CAAE: 73520523.7.0000.0068
Record Dates: First submitted 2024-02-08; First posted 2024-02-29 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-05

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension; Physical Disability; Fragility
Keywords: Pulmonary Endarterectomy Surgery; Six-minute walk test; Short Physical Performance Battery; One-minute sit-to-stand test; Muscular strength; Spirometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational and prospective study is to investigate changes in physical performance, lung function, respiratory and peripheral muscle strength in patients during the postoperative period following pulmonary endarterectomy (PET).

DETAILED DESCRIPTION:
This study aims to investigate the physical changes in patients undergoing pulmonary endarterectomy (PET). It will observe alterations in physical performance, lung function, and muscle strength during the postoperative period. This study, observational and prospective, will include individuals aged ≥18 scheduled, evaluating them preoperatively, post-intensive care unit discharge, before hospital discharge and after six months . Assessments involve tests like the Six-minute walk test, Short Physical Performance Battery, One-minute sit-to-stand test, manovacuometry, dynamometry, spirometry and Clinical Frailty Scale to identify frailty and measure muscle and lung function. The study also aims to explore predictive variables for functional loss during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Both genders
* Elective pulmonary endarterectomy surgery
* Absence of cognitive or peripheral motor impairment that prevents the performance of functional tests in the preoperative period.

Exclusion Criteria:

* Reoperation for any reason
* Presence of cognitive or peripheral motor impairment that prevents the performance of functional tests in the postoperative period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the preoperative period of elective pulmonary endarterectomy susrgery.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
To investigate changes in physical performance measured by Six-Minute Walk Test. | Baseline (one day before the surgery), after the surgery (the day immediately ICU discharge), before the hospital discharge (an average of 20 days) and 6 months after the surgery.
  Measures: the assessment will take place in a flat 30-meter corridor, marked every 1 meter with non-slip flooring, and the patient will be instructed to walk for six minutes as fast as possible.
To investigate changes in physical performance measured by Short Physical Performance Battery (SPPB). | Baseline (one day before the surgery), after the surgery (the day immediately after ICU discharge), before the hospital discharge (an average of 20 days) and 6 months after surgery.
  Measure: global score
To investigate changes in physical performance by 1-minute sit-to-stand test (1-MSTST). | Baseline (one day before the surgery), after the surgery (the day immediately ICU discharge), before the hospital discharge (an average of 20 days) and 6 months after the surgery
  Measure: number of 1-MSTST repetitions.
To investigate changes in peripheral muscle strength. | Baseline (one day before the surgery), after the surgery (the day immediately ICU discharge), before the hospital discharge (an average of 20 days) and 6 months after the surgery
  Measure: hand grip strengh (Kgf).
To investigate changes in respiratory muscle strength: | Baseline (one day before the surgery), after the surgery (the day immediately ICU discharge), before the hospital discharge (an average of 20 days) and 6 months after the surgery
  Measures: manovacuometry (cmH2O)
To investigate changes in lung function test measure by spirometry: | Baseline (one day before the surgery), after the surgery (the day immediately ICU discharge), before the hospital discharge (an average of 20 days) and 6 months after the surgery
To investigate frailty by Clinical Frailty Scale (CFS) | Baseline (one day before the surgery), after the surgery (the day immediately ICU discharge), before the hospital discharge (an average of 20 days) and 6 months after the surgery
  The minimal value is 1 and the maximal is 9 in which the lowest scores mean worse outcomes.

SECONDARY OUTCOMES:
To explore potential preoperative and immediate postoperative risk factors as predictors of functional loss. | Baseline (one day before the surgery) during the immediate postoperative period.
  Measures: Occurrence of comorbidities and clinical variables associated with functional decline.
To investigate changes in hemodynamic and respiratory variables during the funcional tests. | Immediateley before and after each functional test.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael M Ianotti, PT, Principal Investigator — Instituto do Coração - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo
Locations (1):
- Instituto do Coração - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil